CLINICAL TRIAL: NCT06876155
Title: Prospective, Randomized Comparative Study Between an Anesthesiological, Ultrasound-guided, and a Laparoscopic, Landmark-based Application of a "Transversus Abdominis Plane (TAP) Block" Based on Postoperative Pain Perception, Postoperative Analgesic Requirement, and Procedure Duration
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sana Klinikum Offenbach (Other)
Responsible Party: Principal Investigator, Haitham Mutlak, Prof. Dr., Sana Klinikum Offenbach
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-3472-evBO
Record Dates: First submitted 2025-03-04; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Regional Anaesthesia; Transversus Abdominis Plane Block
Keywords: prospective randomised trial; 4 quadrant TAP-Block; Transversus Abdominis Plane Block; ultrasound-guided Transversus Abdominis Plane Block; laparoscopic, landmark-based Transversus Abdominis Plane Block

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: anaesthesiologically performed, ultrasound-guided, dual (lateral & subcostal) TAP block (Active Comparator): The anaesthesiologically performed, ultrasound-guided, 4 quadrant-TAP block ( a combination of a lateral with a subcostal TAP block bilaterally) is performed by an experienced anaesthetist after induction of anaesthesia and before the start of the surgery. A total of 4 punctures are performed. Injection of a total of 60 ml ropivacaine 0.2% into the target compartment (2x 20 ml laterally, 2x 10 ml subcostally)
  Interventions: Procedure: Arm 1: The anaesthesiologically performed, ultrasound-guided, 4 quadrant-TAP block ( a combination of a lateral with a subcostal TAP block bilaterally)
- Arm 2: surgically performed, laparoscopic landmark-based TAP block (Active Comparator): The surgically performed, laparoscopic landmark-based assisted TAP block is performed intraoperatively by the surgeon after the establishment of the pneumoperitoneum and the insertion of the camera. The puncture needle is inserted from the outside under continuous laparoscopic visualization. The spread of the local anaesthetic is continuously visually monitored and should cause a bulging of M. transversus abdominis inward, away from M. obliquus internus ('Doyle's Bulge').
  Injection of a total of 6 x 10 ml = 60 ml ropivacaine 0.2% into the target compartment (at 3 defined puncture sides bilaterally: at the anterior axillary line at 2 different, fixed heights and at the midclavicular line subcostally)
  Interventions: Procedure: Arm2: The surgically performed, laparoscopic landmark-based assisted TAP block

INTERVENTIONS:
Procedure: Arm 1: The anaesthesiologically performed, ultrasound-guided, 4 quadrant-TAP block ( a combination of a lateral with a subcostal TAP block bilaterally) — Injection of a total of 60 ml ropivacaine 0.2% into the target compartment (2x 20 ml laterally, 2x 10 ml subcostally)
  Arms: Arm 1: anaesthesiologically performed, ultrasound-guided, dual (lateral & subcostal) TAP block
Procedure: Arm2: The surgically performed, laparoscopic landmark-based assisted TAP block — Injection of a total of 6 x 10 ml = 60 ml ropivacaine 0.2% into the target compartment (at 3 defined puncture sides bilaterally: at the anterior axillary line at 2 different, fixed heights and at the midclavicular line subcostally)
  Arms: Arm 2: surgically performed, laparoscopic landmark-based TAP block

SUMMARY:
The Transversus Abdominis Plane Block (TAP) has become one of the most established and frequently performed trunk wall blocks for perioperative analgesia in abdominal surgical procedures. The TAP-Block can be performed by both surgeons and anaesthetists.

The goal of this prospective, randomized study is to compare an anesthesiological, ultrasound-guided "Transversus Abdominis Plane (TAP) Block" with a laparoscopic, landmark-based "Transversus Abdominis Plane (TAP) Block"

The main questions it aims to answer are:

Primary Hypothesis: There are no differences in postoperative pain perception and analgesic requirements between the anaesthesiological ultrasound-guided and the surgical laparoscopic landmark-based TAP block

Secondary Hypothesis: There are no significant differences in the duration of the procedure between the anaesthesiological, ultrasound-guided and the surgical laparoscopic landmark-based TAP block.

DETAILED DESCRIPTION:
The Transversus Abdominis Plane Block (TAP) has become one of the most established and frequently performed trunk wall blocks for perioperative analgesia in abdominal surgical procedures. A TAP block is a so-called trunk wall block where a targeted injection of high volumes of local anesthetics is made into a space between two muscle fascias, the so-called inter-fascial space. In this inter-fascial space, the cutaneous nerve branches of various anterior rami of the spinal nerves run and innervate somatosensory in the respective dermatome, skin, soft tissues, and bones, as well as the outer layers of the pleura and peritoneum. Specifically, in a TAP block, the nerve fibers of the spinal nerves from the spinal segments Th6 to L1 can be anaesthetized by applying local anaesthetics between the Musculus obliquus internus abdominis and the Musculus transversus abdominis. The block produces somatic analgesia of the skin, muscles, and bony structures. Visceral analgesia of the internal organs is not achieved. Therefore, the TAP block mainly has an indication within the framework of a multimodal pain concept to save central and peripheral analgesics.

In the literature, it is shown that especially laparoscopic procedures benefit from a TAP block in terms of reducing postoperative reported pain intensity and reducing postoperative opioid requirements. Compared to simple wound infiltration with a local anaesthetic or simple local anaesthesia of the trocar insertion sites in a laparoscopy, the TAP block has been shown to be a more effective method in multiple studies.

The so-called Transversus Abdominis Plane compartment can be reached using various approaches (posterior, lateral, subcostal) and puncture techniques (landmark-based, ultrasound-guided, and surgical). A lateral approach is used primarily for analgesia in lower abdominal surgery (e.g., inguinal hernia repair). A subcostal approach is used primarily for analgesia in upper abdominal/supraumbilical surgery (e.g., cholecystectomy). A dual TAP block or '4 quadrant block,' the combination of a lateral with subcostal TAP block, could achieve better abdominal distribution of the local anaesthetic and more complete analgesia for the lower (T10-T12) and upper (T6-T9) abdomen.

The goal of this monocentric, prospective, randomised study is to compare an anesthesiological, ultrasound-guided "Transversus Abdominis Plane (TAP) Block" with a laparoscopic, landmark-based "Transversus Abdominis Plane (TAP) Block" in two parallel study arms.

Anaesthesia Induction and maintenance in both groups are standardised and similar.

The main questions to answer are:

Primary Hypothesis: There are no differences in postoperative pain perception and analgesic requirements between the anaesthesiological ultrasound-guided and the surgical laparoscopic landmark-based TAP block

Secondary Hypothesis: There are no significant differences in the duration of the procedure between the anaesthesiological, ultrasound-guided and the surgical laparoscopic landmark-based TAP block.

A sample size calculation was performed before study start. The hypotheses will be verified by suitable statistical analysis. The randomization process is performed preoperatively using a closed envelope ('Sealed Envelope') that assigns a patient to one of the two intervention groups.

ELIGIBILITY:
Inclusion Criteria:

* Consent of the adult patient
* Elective laparoscopic-assisted colorectal surgery, elective laparoscopic cholecystectomy, or elective laparoscopic fundoplication

Exclusion Criteria:

* Lack of patient consent
* Pregnancy and breastfeeding
* Allergies to local anaesthetics used
* Infections at the puncture sites
* History of complex abdominal wall reconstruction
* Chronic pain syndrome
* Fibromyalgia
* Chronic opioid use
* Chronic alcohol abuse
* Chronic drug abuse (THC, amphetamines, cocaine, etc.)
* Psychiatric preconditions (depression, schizophrenia, etc.)
* Patients with impaired consciousness, communication, or cognitive function
* Diagnosed coagulopathies (e.g., platelet count <80,000/µL, PTT/aPTT- prolongation >1.5 upper normal value)
* Therapeutic anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Assessment of the postoperative pain perception using the NRS pain scale | First 24 hours postoperatively
  Standardized pain assessments postoperatively are conducted by the in-house anaesthesiological pain service using a standardized pain form (which consists of a NRS Scoring in rest and at motion at fixed times [1 hour, 2 hours, 6 hours, 12 hours, 24 hours]).
  The anaesthesiological pain service is blinded to the procedure performed.
Assessment of the postoperative analgesic requirements/consumption within the first 24 hours after surgery | First 24 hours postoperatively
  An assessment of the cumulative analgesic consumption in the first 24 hrs. postoperatively is conducted by the in-house anaesthesiological pain service. Both total opioid consumption (in mg) and consumption of basic analgetics (e.g. paracetamol, metamizole, etc.)(in mg) are measured.
  The anaesthesiological pain service is blinded to the procedure performed.

SECONDARY OUTCOMES:
Duration of the TAP block procedure | perioperatively
  Duration of the TAP block procedure, defined as the time from the first needle introduction to the completed application of the total amount of the local anaesthetic (in minutes).

OTHER OUTCOMES:
PONV-Incidence | First 24 hours postoperatively
  The incidence of PONV
Duration of the patient stay in the recovery room | First 24 hours postoperatively
  Total amounts of minutes that the patient was monitored in the recovery room before dismissal to normal ward
Complications | First 24 hours postoperatively
  Incidence of complications

CONTACTS AND LOCATIONS:
Overall Officials: Prof.Dr. H. Mutlak, Principal Investigator — Department of Anaesthesiology, Intensive Care Medicine, and Pain Therapy at the Sana Klinikum Offenbach
Locations (1):
- Director of the Department of Anaesthesiology, Intensive Care Medicine, and Pain Therapy at the Sana Klinikum Offenbach, Offenbach, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No